CLINICAL TRIAL: NCT00949637
Title: A Site-Randomized Controlled Trial for Health Promotion in Girl Scouts: Healthier Troops in a SNAP
Brief Title: Scouting Nutrition and Activity Program
Acronym: SNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: The Sunflower Foundation (Unknown)
Responsible Party: Principal Investigator, Richard R. Rosenkranz, Assistant Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SF SNAP y1
Record Dates: First submitted 2009-07-21; First posted 2009-07-30 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: obesity prevention; girl scouts; physical activity; family meals; fruits and vegetables; health promotion
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scouting curricular implementation (Experimental): Intervention group will receive a curriculum based on social cognitive theory, wherein children will be taught skills in a supportive environment to improve their self efficacy and proxy efficacy toward eating healthful meals and being physically active with a parent. Troop leaders and parents will provide support, and help girls to create healthy opportunities in the home environment. Simultaneously, girls will be taught skills to improve the family mealtime environment, to bolster asking skills toward healthy behavior, to self-monitor healthy behavior, and to set goals for healthy behavior.
  Interventions: Behavioral: Scouting Nutrition and Activity Program
- Standard-care attentional control (Active Comparator): Control troops complete usual troop meeting activities. Control troops receive equal observation time, equal pretest and posttest assessment, and equal study scrutiny.
  Interventions: Behavioral: Standard-care attentional control

INTERVENTIONS:
Behavioral: Scouting Nutrition and Activity Program — Intervention group will receive a curriculum based on social cognitive theory, wherein children will be taught skills in a supportive environment to improve their self efficacy and proxy efficacy toward eating healthful meals and being physically active with a parent. Troop leaders and parents will provide support, and help girls to create healthy opportunities in the home environment. Simultaneously, girls will be taught skills to improve the family mealtime environment, to bolster asking skills toward healthy behavior, to self-monitor healthy behavior, and to set goals for healthy behavior.
  Other Names: SNAP
  Arms: Scouting curricular implementation
Behavioral: Standard-care attentional control — Control troops complete usual troop meeting activities. Control troops receive equal observation time, equal pretest and posttest assessment, and equal study scrutiny.
  Other Names: Control
  Arms: Standard-care attentional control

SUMMARY:
The purpose of the study was to evaluate the effectiveness of an intervention designed to prevent obesity by improving the environmental characteristics of Girl Scouts troop meetings.

DETAILED DESCRIPTION:
Girls and parents affiliated with Girl Scouts Juniors programs completed a questionnaire prior to the beginning of an intervention program, and again after the program. Children responded to previously validated questionnaire items assessing demographics, parent-child connectedness, parent-child physical activity, screen time usage, family meal-time environment, consumption of fruits and vegetables, soda, and fast food. Parents completed a similar questionnaire, assessing demographics, parent-child connectedness, parent-child physical activity, family mealtime environment, parenting style and parenting practices. Children were also assessed on height and weight to characterize their risk for overweight status. Questionnaires and environmental observations were used to assess the effectiveness of an intervention designed to improve the family meal-time environment at home, as well as helping to assess the relationships between parental factors and family health-related behavior.

ELIGIBILITY:
Inclusion Criteria:

* Girls had to be attending members of Girl Scouts in one of our included troops.
* The troop needed to be a registered Girl Scouts Juniors troop, consisting of girls primarily in the 4th and 5th grades.
* To be officially registered, the troop leaders were required to complete Girl Scout leader training and pass a criminal background check.
* To be included, the troops also needed to meet at least twice per month, have meeting facilities capable of allowing physical activity and food preparation.
* Also, troops needed to have initial agreement of leaders and parents for the troop to participate in a research study.

Exclusion Criteria:

* An inability to speak or read English.
* Troops not primarily composed of Girl Scouts Juniors, not regularly meeting during the study period, or not having leader and parental consensus approval for troop participation.

Ages: 8 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Body mass index percentile ranking | 5 months

SECONDARY OUTCOMES:
Obesity-related behaviors | 5 months
Troop environmental encouragement and opportunities for healthful eating and physical activity | continuous

CONTACTS AND LOCATIONS:
Overall Officials: Richard R. Rosenkranz, PhD, Principal Investigator — Kansas State University
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

REFERENCES:
- [Result] Rosenkranz RR, Behrens TK, Dzewaltowski DA. A group-randomized controlled trial for health promotion in Girl Scouts: healthier troops in a SNAP (Scouting Nutrition & Activity Program). BMC Public Health. 2010 Feb 19;10:81. doi: 10.1186/1471-2458-10-81. PMID 20170502